CLINICAL TRIAL: NCT02961322
Title: Medico-economic Study of the Lobo-isthmectomy Assisted Robot
Acronym: LIRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough inclusions
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9657
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Lobo-isthmectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lobo isthmectomy (Experimental)
  Interventions: Other: lobo-isthmectomy assisted robot

INTERVENTIONS:
Other: lobo-isthmectomy assisted robot

SUMMARY:
This is a study of health economics longitudinal cohort on the evaluation of direct medical cost of a surgical technique based on the use of an innovative device (the da Vinci® surgical robot Si) and its comprehensive care.

DETAILED DESCRIPTION:
Over 50,000 thyroidectomies are performed each year in France. The externally surgery produces satisfactory results, but it nevertheless remains a risk of complications in the order of 10 to 20%. Moreover, the patients operated by traditional externally have a basi-cervical visible scar which is a major concern for many of them. The team of Montpellier University Hospital is a pioneer in the use of the technique of endoscopic thyroidectomy under robotic assistance that saves totally cervical scarring for patients, but also decrease the rate of complications. This technique based on the use of the da Vinci robotic system if justified, depending on the manufacturer and the scientific literature, with its minimally invasive character, an amplitude of greater movement than the hand of man, and movements called intuitive that reduce tremors instruments during the operation (Patel 2008). In France and in Europe, there is a growing demand from patients and surgeons to access the surgical technique. An assessment of the real and specific cost of this technique and its overall management is essential in order to assess the financial impact of the introduction of this surgery for our hospitals, or no data is available on this in Literature.

The main objective of this study is to describe the direct medical cost of the treatment of thyroid Lobo-Isthmectomy Robot-Assisted (LIRA) with a follow-up 12 months. The secondary objectives of this research are to determine the rate of laryngeal paralysis, the rate of complications specific to access axillary robot, the size of the incision made for surgery, the number of channel conversion transaxillary assisted robot traditional externally, to assess the satisfaction of each patient over his scar, pain over time, the evolution of potential disorders sensitivity of anterior chest wall, the vocal functional suites and quality of life self-administered questionnaire (Voice handicap Index VHI 10 and Short Forme SF-36), and finally to compare the cost of care by the robot with the average cost of a conventional surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient candidate for thyroid lobectomy or lobo-isthmectomy for benign nodular disease
* normal laryngeal mobility (clinical evaluation by an ENT (Ear-Nose-Throat) Doctor)
* breast cancer absence being supported
* No suspected thyroid cancer
* Nodules size <6cm
* Confirm Benin character nodules by fine needle biopsy made within 6 months prior to patient inclusion
* Patient available for post-operative follow-up of 12 months

Exclusion Criteria:

* Patient participating or having participated in another interventional study in the previous 3 months or exclusion period determined by a previous study
* Patient under guardianship or trusteeship or under judicial protection
* Inability to give informed patient information
* Pregnant women, breastfeeding or parturient
* Contraindications (or incompatible combination therapy) for a necessary treatment in this study
* contraindication to general anesthesia
* Emergencies
* Breast Cancer being supported
* treatment or surgical sentinel node of the planned breast cancer
* thyroid nodule ranked in the ultrasound TIRADS 5 (Thyroid image reporting and data system)
* Fine needle aspiration biopsy with BETHESDA score result 5 and 6
* Plunging Nodule

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
direct medical cost | 12 months

IPD SHARING:
Plan to Share IPD: No